CLINICAL TRIAL: NCT00147121
Title: Rituximab + Standard CHOP (R･S-CHOP) vs Rituximab+ Bi-weekly CHOP (R･Bi-CHOP) RCT(Phase II/III) for Stage III/IV Low-grade B-cell Lymphoma (LowBNHL-RS/BiCHOP-P2/3) (JCOG0203)
Brief Title: Rituximab+Standard CHOP vs Rituximab+Bi-weekly CHOP for Untreated Stage III/IV Low-grade B-cell Lymphoma (JCOG0203)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Haruhiko Fukuda (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor-Investigator, Haruhiko Fukuda, JCOG Data Center, Japan Clinical Oncology Group
Organization: Japan Clinical Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0203; C000000033
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Lymphoma, B-Cell
Keywords: Rituximab; CHOP; Bi-weekly; low-grade B-cell lymphoma; advanced stage; follicular lymphoma; G-CSF; Untreated stage III/IV low-grade B-cell lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Rituximab+Standard CHOP
  Interventions: Drug: Rituximab + Standard CHOP
- 2 (Experimental): Rituximab+bi-Weekly CHOP
  Interventions: Drug: Rituximab + Bi-weekly CHOP

INTERVENTIONS:
Drug: Rituximab + Standard CHOP — Rituximab + Standard CHOP
  Arms: 1
Drug: Rituximab + Bi-weekly CHOP — Rituximab + Bi-weekly CHOP
  Arms: 2

SUMMARY:
To establish standard therapy for patients with advanced-stage low grade B-cell lymphoma

DETAILED DESCRIPTION:
Since currently there is no standard therapy for untreated advanced-stage low-grade B-cell lymphoma, Phase 2/3 study was planned. Comparison(s): An intensified bi-weekly version by shortening the intervals of both rituximab and CHOP therapies using G-CSF, compared to the tri-weekly R-CHOP regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmed, low-grade B-cell lymphoma except mantle cell lymphoma and histologic transformation to DLBCL
2. CD20-positive
3. Ann Arbor CS III or IV
4. Lymphoma cell count in PB≦10,000/mm3
5. 20<=age<=69
6. ECOG PS 0-2
7. Bidimensionally measurable disease >1.5cm in a single dimension by CT scans
8. No prior chemotherapy, radiotherapy, interferon-alfa, or antibody therapy
9. Normal BM, hepatic, renal, cardiac, and pulmonary function
10. Written informed consent

Exclusion Criteria:

1. CNS involvement
2. Glaucoma
3. DM treated by insulin
4. Uncontrollable HT
5. AP, AMI
6. Positive HBs antigen
7. seropositive to HCV
8. seropositive to HIV
9. Interstitial pneumonitis, pulmonary fibrosis, or emphysema
10. Severe infection
11. Liver cirrhosis
12. Double cancer
13. Pregnant or lactating
14. Patients who desire auto PBST after CR
15. Patients treated with major tranquilizer or antidepressant

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2002-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
CR rate (phase II) | during the study conduct
PFS (phase III) | during the study conduct

SECONDARY OUTCOMES:
ORR, PFS, OS, Safety (phase II) | during the study conduct
OS, Safety (phase III) | during the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, M.D.,Ph.D., Study Chair — National Cancer Center Hospital
Locations (45):
- Japan (45):
  - Aichi Medical University, Aichi-gun,Nagakute,Yazako,Karimata,21, Aichi-ken
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Nagoya City University Hospital, Nagoya,Mizuho-ku,Mizuho-cho,Kawasumi,1, Aichi-ken
  - Nagoya University School of Medicine, Nagoya,Showa-ku, Tsurumai-cho,65, Aichi-ken
  - Nagoya Daini Red Cross Hospital, Nagoya,Showa-ku,Myoken-cho,2-9, Aichi-ken
  - Nagoya Medical Center, Nagoya,Naka-ku,Sannomaru,4-1-1, Aich
  - Akita University School of Medicine, Akita,Hondo,1-1-1, Akita
  - Chiba Cancer Center Hospital, Chiba,Chuo-ku,Nitona-cho,666-2, Chiba
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - Ehime University Hospital, Shitsukawa,Toon, Ehime
  - University of Fukui Hospital, Yoshida-gun,Matsuoka,Shimoaizuki,23-3, Fukui
  - School of Medicine,Fukuoka University, Fukuoka,Jonan-ku,Nanakuma,7-45-1, Fukuoka
  - National Kyushu Cancer Center, Fukuoka,Minami-ku,Notame,3-1-1, Fukuoka
  - National Hospital Organization Kyusyu Medical Center, FukuokaChuo-ku,Jigyohama,1-8-1, Fukuoka
  - University of Occupational and Environmental Health, Kitakyushu,Yahatanishi-ku,Iseigaoka,1-1, Fukuoka
  - Ohta Nishinouchi Hospital, Kohriyama,Nishinouchi,2-5-20, Fukushima
  - Gunma University, Maebashi,Showa,3-39-15, Gunma
  - Sapporo Hokuyu Hospital, Sapporo,Shiroishi-ku,Higashi-sapporo,6-5-1, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo,Shiroishi-ku,Kikusui,4-2-3-54, Hokkaido
  - Kanazawa Medical University, Kahoku-gun,Uchinada-machi,Daigaku,1-1, Ishikawa-ken
  - Imamura Bun-in Hospital, Kagoshima,Kamoikeshinmachi,11-23, Kagoshima-ken
  - Kagoshima University,Faculty of Medicine, Kagoshima,Sakuragaoka,8-35-1, Kagoshima-ken
  - Tokai University School of Medicine, Isehara,Shimokasuya,143, Kanagawa
  - St.Marianna University School of Medicine,Yokohama City Seibu Hospital, Yokohama,Asahi-ku,Yasashi-cho,1197-1, Kanagawa
  - Kumamoto University Medical School, Kumamoto,Honjo,1-1-1, Kumamoto
  - NHO Kumamoto Medical Center, Kumamoto,Ninomaru,1-5, Kumamoto
  - Kyoto Prefectural University of Medicine, Kyoto,Kamigyo-ku,Kawaramachi-Hirokoji,465, Kyoto
  - Mie University School of Medicine, Tsu,Edobashi,2-174, Mie-ken
  - Tohoku University Hospital, Sendai,Aoba-ku,Seiryo-machi,1-1, Miyagi
  - Nagasaki University Hospital, Nagasaki,Sakamoto,1-7-1, Nagasaki
  - Nagasaki Medical Center, Oomura,Kubara,2-1001-1, Nagasaki
  - Sasebo City General Hospital, Sasebo,Hirasemachi,9-3, Nagasaki
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Oita Prefectural Hospital, Oita,Bunyo,476, Oita Prefecture
  - Faculty of Medicine,University of Ryukyus, Nakagami,Nishihara,Uehara,207, Okinawa
  - Faculty of Medicine, Saga University, Saga,Nabeshima,5-1-1, Saga-ken
  - Saitama Cancer Center, Kita-adachi,Ina,Komuro,818, Saitama
  - Shiga Medical Center for Adults, Moriyama,Moriyama,5-4-30, Shiga
  - Hamamatsu University School of Medicine, Hamamatsu,Handayama,1-20-1, Shizuoka
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku,Honkomagome,3-18-22, Tokyo
  - National Cancer Center Hospital, Chuo-kum,Tsukiji, 5-1-1, Tokyo
  - Jikei University,Daisan Hospital, Komae,Izumihoncho,4-11-1, Tokyo
  - Jikei University Hospital, Minato-ku,Nishishinbashi,3-25-8, Tokyo
  - Kyorin University School of Medicine, Mitaka,Shinkawa,6-20-2, Tokyo
  - Tokyo Medical University, Shinjuku-ku,Nishi-shinjuku,6-7-1, Tokyo

REFERENCES:
- [Derived] Watanabe T, Tobinai K, Wakabayashi M, Maruyama D, Yamamoto K, Kubota N, Shimada K, Asagoe K, Yamaguchi M, Ando K, Ogura M, Kuroda J, Suehiro Y, Matsuno Y, Tsukasaki K, Nagai H. R-CHOP treatment for patients with advanced follicular lymphoma: Over 15-year follow-up of JCOG0203. Br J Haematol. 2024 Mar;204(3):849-860. doi: 10.1111/bjh.19213. Epub 2023 Nov 23. PMID 37996986
- [Derived] Watanabe T, Tobinai K, Wakabayashi M, Morishima Y, Kobayashi H, Kinoshita T, Suzuki T, Yamaguchi M, Ando K, Ogura M, Taniwaki M, Uike N, Yoshino T, Nawano S, Terauchi T, Hotta T, Nagai H, Tsukasaki K; JCOG0203 Collaborators. Outcomes after R-CHOP in patients with newly diagnosed advanced follicular lymphoma: a 10-year follow-up analysis of the JCOG0203 trial. Lancet Haematol. 2018 Nov;5(11):e520-e531. doi: 10.1016/S2352-3026(18)30155-8. PMID 30389034
- [Derived] Watanabe T, Tobinai K, Shibata T, Tsukasaki K, Morishima Y, Maseki N, Kinoshita T, Suzuki T, Yamaguchi M, Ando K, Ogura M, Taniwaki M, Uike N, Takeuchi K, Nawano S, Terauchi T, Hotta T. Phase II/III study of R-CHOP-21 versus R-CHOP-14 for untreated indolent B-cell non-Hodgkin's lymphoma: JCOG 0203 trial. J Clin Oncol. 2011 Oct 20;29(30):3990-8. doi: 10.1200/JCO.2011.34.8508. Epub 2011 Sep 19. PMID 21931035
- See also: Related Info — http://www.jcog.jp/